CLINICAL TRIAL: NCT03015961
Title: A Multicenter, Randomized, Double-Blind, Controlled Study of EXPAREL for Postsurgical Pain Management in Subjects Undergoing Open Lumbar Spinal Fusion Surgery
Brief Title: Phase 4, Controlled Study in Adult Subjects Undergoing Primary, 1-2 Level, Open Lumbar Spinal Fusion Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-409
Record Dates: First submitted 2016-11-14; First posted 2017-01-10 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain Management
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EXPAREL admixed with bupivacaine HCl (Active Comparator): EXPAREL 266 mg + bupivacaine HCl
  Interventions: Drug: EXPAREL and bupivacaine HCl
- Bupivacaine HCl (Placebo Comparator): Bupivacaine HCl
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: EXPAREL and bupivacaine HCl — Drug: EXPAREL EXPAREL and bupivacaine HCl
  Other Name: bupivacaine liposome injectable suspension Drug: Bupivacaine Single dose of bupivacaine HCl 0.5%
  Other Name: bupivacaine HCl
  Arms: EXPAREL admixed with bupivacaine HCl
Drug: Bupivacaine HCl — Drug: Bupivacaine Single dose of bupivacaine HCl 0.5%
  Other Name: bupivacaine HCl
  Arms: Bupivacaine HCl

SUMMARY:
Primary Objective: The primary objective of this study is to compare postsurgical pain control following local infiltration analgesia (LIA) with EXPAREL admixed with bupivacaine HCl versus LIA with bupivacaine HCl in adult subjects undergoing open lumbar posterior spinal fusion surgery.

Secondary Objectives: The secondary objectives of this study are to compare additional efficacy, safety, and health economic outcomes following LIA with EXPAREL admixed with bupivacaine HCl versus LIA with bupivacaine HCl in adult subjects undergoing open lumbar posterior spinal fusion surgery.

DETAILED DESCRIPTION:
This is a Phase 4, multicenter, randomized, double-blind, controlled study in 38 adult subjects undergoing primary, 1-2 level, open lumbar spinal fusion surgery under general anesthesia.

Subjects will be screened within 30 days prior to study drug administration and at least one day prior to surgery. During the screening visit, subjects will be assessed for past or present neurologic, cardiac, and general medical conditions that in the opinion of the Investigator would preclude them from study participation. After the informed consent form (ICF) is signed, a medical history, surgical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, select clinical laboratory evaluations, urine drug screen, alcohol breath test, and urine pregnancy test for women of childbearing potential will be conducted. Study drug, approximately 1-2 mL every 1.0-1.5 cm, will be administered using 20- or 22-gauge needles prior to wound closure.

Administration Instructions/Procedures

Study drug should be injected in the prescribed locations based on the areas of highest nerve density. Study drug will be administered using syringes with 20- or 22-gauge needles prior to wound closure. The Investigator must document the size of the incision. Each infiltration site should be spaced 1.0-1.5 cm apart and should deliver approximately 1-2 mL into both deep and superficial areas (para-spinous fascia, muscle, and subcutaneous layers). Total volume administered will be depended on the number of levels of dissection, as described below. Following infiltration, the tissue should visibly expand with minimal leakage.

Total Volume of Expansion

The Investigator must document the total volume used for each surgery.

1. Level Procedures Group 1: EXPAREL 266 mg in 20 mL + bupivacaine HCl 0.5% in 20 mL + 20 mL normal saline = total volume of 60 mL Group 2: Bupivacaine HCl 0.5% in 20 mL + 40 mL normal saline = total volume of 60 mL
2. Level Procedures Group 1: EXPAREL 266 mg in 20 mL + bupivacaine HCl 0.5% in 20 mL + 50 mL normal saline = total volume of 90 mL Group 2: Bupivacaine HCl 0.5% in 20 mL + 70 mL normal saline = total volume of 90 mL

Drains may be used at the surgeon's discretion. In addition to LIA, all study participants will receive a standardized approach for managing postsurgical pain that includes a scheduled multimodal pain regimen including adjunctive analgesics, non-steroidal anti-inflammatory drugs (NSAIDs). Rescue analgesics will be available as needed.

Postsurgical clinical assessments will include pain intensity scores using a 10-cm visual analog scale (VAS) (see Appendix 1); overall benefit of analgesia score (OBAS) questionnaire (see Appendix 2); total postsurgical opioid consumption; predefined opioid-related AEs; and nurse's satisfaction with overall analgesia (see Appendix 3).

Adverse events will be recorded from the time the ICF is signed through Day 30. If a cardiac AE (e.g., chest pain [angina, myocardial infarction], abnormal/irregular heart rate [bradycardia, tachycardia, extrasystoles], or shortness of breath), neurological AE (e.g., altered mental status/altered sensorium, dizziness, dysarthria, hyperesthesia, metallic taste, peroral numbness, seizure, tinnitus, tremors, visual disturbance, muscular twitching or rigidity beyond 72 hours postdose, or tingling/paresthesia beyond 72 hours postdose), or serious AE (SAE) occurs during the study a 12-lead ECG, vital signs, and any appropriate clinical laboratory tests should be conducted.

Postsurgical health economic outcome assessments will include hospital length of stay (LOS), use of skilled nursing facility, hospital readmissions, and use of other health services following discharge (phone calls related to postsurgical pain, unscheduled visits related to postsurgical pain, and visits to emergency department) through Day 30.

A follow-up visit will be scheduled for all subjects on postsurgical Day 14. A follow-up phone call will be made on Day 30 to all subjects who received study drug to assess for adverse events (AEs).

Number of Subjects (Planned):

Approximately 194 subjects are planned for enrollment in this study in order to have at least 184 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age at screening.
2. Primary surgical indication is lumbar pain, radiculopathy, disc degeneration, disc herniation, foraminal stenosis, or 1-2 level spondylolisthesis or deformity.
3. Scheduled to undergo primary, 1-2 level, open lumbar spinal fusion surgery under general anesthesia.
4. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
5. Female subjects must be surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, or transdermal, contraceptive approved by the FDA for greater than 2 months prior to screening. All women of childbearing potential (ie, premenopausal without permanent sterilization) must commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study.
6. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
2. Serious spinal conditions (to include cauda equina syndrome, infection, tumor, fracture, or severe osteoporosis [ie, if taking Bisphosphonate or TNF-α blockers]).
3. Planned anterior or lateral incisions
4. Previous spinal surgery at the same level other than microdiscectomy or hemilaminectomy (eg, bi-lateral laminectomy, fusion).
5. Planned concurrent surgical procedure.
6. Identification of a dural tear during surgery will be an intra-operative exclusion unless it is well repaired (no evidence of cerebrospinal fluid [CSF] leak with Valsalva and no plan to restrict activity post-operatively). Any injury to the nerve root occurring during surgery will also be considered an intra-operative exclusion.
7. Concurrent painful physical condition that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the spinal surgery and which may confound the postsurgical assessments.
8. Comorbidity impacting current physical function or Investigator opinion that it may impact postsurgical rehabilitation.
9. Allergy, hypersensitivity, or contraindication to any of the study medications (ie, bupivacaine, oxycodone, morphine, hydromorphone, gabapentin, acetaminophen, or cyclobenzaprine) for which an alternative medication is not provided in the protocol.
10. Use of any of the following medications within the times specified before surgery: long-acting opioid medication (eg, morphine including MS Contin®, hydromorphone [Dilaudid®], oxycodone [Oxycontin®], methadone) daily for more than 3 months duration or within 3 days of surgery. Patients receiving short-acting opioids or NSAIDs should be at a steady or plateau dose. Such patients should require or receive no more than 40 mg morphine (oral) equivalents (eg, approximately 5 mg oxycodone) within 24 hours of surgery.
11. Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, he or she must be on a stable dose for at least 1 month prior to study drug administration.
12. Current use of systemic glucocorticosteroids within 1 month of enrollment in this study.
13. Use of dexmedetomidine HCl (Precedex®) within 3 days of study drug administration.
14. History of coronary or vascular stent placed within the past 3 months (may be extended to 1 year if medically indicated per physician discretion).
15. Have been treated for a deep vein thrombosis, pulmonary embolism, myocardial infarction, or ischemic stroke within the past 6 months (may be extended to 1 year if medically indicated per physician discretion).
16. Severely impaired renal (eg, serum creatinine clearance ≤ 30) or hepatic function (eg, serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN] or serum alanine aminotransferase [ALT] level >3 x ULN).
17. Any neurologic or psychiatric disorder that might impact postsurgical pain or interfere with study assessments.
18. Malignancy in the last 2 years, per physician discretion.
19. History of misuse, abuse, or dependence on opioid analgesics, other prescription drugs, illicit drugs, or alcohol as defined in DSM-IV. Dependence or chronic opioid use will be defined as use of more than 30 morphine equivalents per day during the prior 90 days.
20. Failure to pass the alcohol breath test or urine drug screen positive for illicit drugs.
21. Body weight <50 kg (110 pounds) or a body mass index >44 kg/m2.
22. Subjects receiving Worker's compensation for a disability or who are involved in litigation.
23. Previous participation in an EXPAREL study.
24. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - OrthoArizona, Gilbert, Arizona
  - St. Joseph's Hospital, Phoenix, Arizona
  - UC Davis, Sacramento, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beaumont Health, Troy, Michigan
  - Washington Univ, St Louis, Missouri
  - Icahn School of Medicine, New York, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Ohio State Univ, Columbus, Ohio
  - Thomas Jefferson University of Neurosurgery, Philadelphia, Pennsylvania
  - Central Texas Spine Institute, Austin, Texas
  - Baylor Scott & White, Temple, Texas
  - Univ of Virginia, Charlottesville, Virginia
  - Colonial Orthopaedics, Colonial Heights, Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February 21, 2017 and October 30, 2017 at 15 sites in the United States. The study was terminated due to low enrollment.
Groups:
- EXPAREL Admixed With Bupivacaine HCl: Local infiltration analgesia with EXPAREL (bupivacaine liposome injectable suspension) 266 mg/20 mL admixed with bupivacaine HCl 0.5% 20 mL and expanded with 20 mL (1-level procedures) or 50 mL (2-level procedures) normal saline
- Bupivacaine HCl: Local infiltration analgesia with bupivacaine hydrochloride (HCl) 0.5% 20 mL expanded with 40 mL (1-level procedures) or 70 mL (2-level procedures) normal saline
Period: Overall Study
Arm/Group | EXPAREL Admixed With Bupivacaine HCl | Bupivacaine HCl
Started | 18 | 20
Completed | 18 | 18
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized subjects. The study was terminated; no efficacy outcomes were analyzed.
Groups:
- Bupivacaine HCl: Local infiltration analgesia with bupivacaine HCl 0.5% 20 mL expanded with 40 mL (1-level procedures) or 70 mL (2-level procedures) normal saline
- Total: Total of all reporting groups
Arm/Group | EXPAREL Admixed With Bupivacaine HCl | Bupivacaine HCl | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: year] | 57.3 (12.13) | 61.6 (9.33) | 59.5 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Visual Analog Scale (VAS) Pain Intensity Scores From 0 to 72 Hours
Description: AUC of VAS pain intensity scores from 0 to 72 hours postsurgery. Visual Analog Scale (VAS) is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now." AUC curve is derived using the trapezoidal rule (see formula below) on the pain scores. AUC start with the first pain assessment obtained after surgery and use all subsequent pain assessments up to 72 hours post-surgery. (Where pi is the VAS pain score at time i and ti is the time, in hours, from end of surgery. Note t1 is pain score collected after surgery.)
Time Frame: 0-72 hours
Measure: Mean (Full Range); unit: score on a scale*hours
Arm/Group | EXPAREL Admixed With Bupivacaine HCl | Bupivacaine HCl
Number analyzed (Participants) | 18 | 20
score on a scale*hours | 342.8 [1 to 624] | 369.0 [96 to 718]

2. Other Pre Specified Outcome: Percentage of Opioid-Free Patients
Description: Percentage of opioid-free patients through 24, 48 and 72 hours post-surgery
Time Frame: 0-24, 0-48, 0-72 hours
Measure: Number; unit: percentage of opioid-free patients
Arm/Group | EXPAREL Admixed With Bupivacaine HCl | Bupivacaine HCl
Number analyzed (Participants) | 18 | 20
percentage of opioid-free patients
  0-24 hours | 11.11 | 11.11
  0-48 hours | 11.11 | 5.56
  0-72 hours | 11.11 | 5.56

3. Other Pre Specified Outcome: Area Under the Curve (AUC) of the Visual Analog Scale (VAS) Pain Intensity Scores From 24-48 and 48-72 Hours Postsurgery
Description: AUC of the VAS pain intensity scores from 24-48 and 48-72 hours postsurgery. Visual Analog Scale (VAS) is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now." AUC from 24-48 hours start with the pain assessment obtained at 24 hours post-surgery and use all subsequent pain assessments up to 48 hours post-surgery. AUC from 48-72 hours start with the pain assessment obtained at 48 hours post-surgery and use all subsequent pain assessments up to 72 hours post-surgery. (Where pi is the VAS pain score at time i and ti is the time, in hours, from end of surgery.)
Time Frame: 24-48 hours, 48-72 hours
Measure: Mean (Full Range); unit: score on a scale*hours
Arm/Group | EXPAREL Admixed With Bupivacaine HCl | Bupivacaine HCl
Number analyzed (Participants) | 18 | 20
score on a scale*hours
  24-48 hours | 97.3 [0 to 185] | 98.1 [14 to 225]
  48-72 hours | 86.8 [0 to 187] | 90.6 [8 to 162]

4. Other Pre Specified Outcome: Total Opioid Consumption Through 48 Hours Postsurgery
Description: Total Opioid Consumption Through 48 Hours Postsurgery
Time Frame: 0-48 hours
Measure: Mean (Standard Deviation); unit: MED, mg
Arm/Group | EXPAREL Admixed With Bupivacaine HCl | Bupivacaine HCl
Number analyzed (Participants) | 18 | 20
MED, mg | 103.6 (101.55) | 90.8 (100.58)

ADVERSE EVENTS:
Time Frame: From the time informed consent form is signed to Day 30
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality. Serious AEs were defined as per clinicaltrials.gov.
Arm/Group | EXPAREL Admixed With Bupivacaine HCl | Bupivacaine HCl
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/20
Other Adverse Events (participants affected / at risk) | 11/18 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL Admixed With Bupivacaine HCl (N=18) | Bupivacaine HCl (N=20)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL Admixed With Bupivacaine HCl (N=18) | Bupivacaine HCl (N=20)
Dizziness (Nervous system disorders) | 0 | 4
Radiculopathy (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Incision site pain (Injury, poisoning and procedural complications) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Hypotension (Vascular disorders) | 0 | 3
Urinary tract infection (Infections and infestations) | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 1
Agitation postoperative (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Pedal pulse decreased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Facial spasm (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to low enrollment; small sample sizes make data interpretation difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT03015961/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03015961/SAP_001.pdf